CLINICAL TRIAL: NCT04749316
Title: Transcutaneous Electric Nerve Stimulation on Acupoints (Acu-TENS) for the Treatment of Faecal Incontinence: a Prospective, Randomised, Sham-controlled Trial.
Brief Title: Acs-Tens Treatment for Faecal Incontinence: a RCT With Sham-controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Tony Wing Chung Mak, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMRF13140421
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Faecal Incontinence; Faecal Incontinence With Faecal Urgency; Neuromodulation; Transcutaneous Electric Nerve Stimulation; Acupuncture Points
Keywords: Faecal incontinence; Faecal urgency; Neuromodulation; Transcutaneous Electric Nerve Stimulation; Acupuncture
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Intervention Model Description: Acutens treatment for faecal incontinence vs sham
Who Masked: Participant, Outcomes Assessor
Masking Description: participant will not be told on which treatment arm are in. Outcome assessors will be blinded on participants' treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AcuTENS (Experimental): Patients treated with TENS over Acupuncture points for faecal incontinence
  Interventions: Procedure: AcuTENS
- Sham (Sham Comparator): Sham treatment arm with no electrical stimulations over acupuncture points
  Interventions: Procedure: AcuTENS

INTERVENTIONS:
Procedure: AcuTENS — Stimulation of acupuncture points with TENS machine

SUMMARY:
This study assess the effectiveness on AcuTENS on the treatment of faecal incontinence

DETAILED DESCRIPTION:
Faecal incontinence (FI) is the involuntary loss of flatus, liquid or solid stool per rectum. Owing to the emotional stress and the psychosocial stigma surrounding this problem, it is under-reported by patients.

Conservative management of FI involves lifestyle, medical adjustments and pelvic floor sphincter training. If conservative treatment fails, surgical options such as sphincter repair, sacral nerve stimulation (SNM) and percutaneous tibial nerve stimulation (PTNS) can be reformed. SNM and PTNS involve application of nervous electrical stimulation (neuromodulation) with significant improvement of symptoms. The positions of electrical stimuli are also very similar to acupuncture sites (acupoints) used in Traditional Chinese Medicine for the treatment of faecal incontinence. However, disadvantage of these methods are; 1) they are invasive and may cause complications such as pain, infection and bleeding and; 2) the devices for each SNM device can be costly.

Transcutaneous Electrical Nerve Stimulation (TENS) is non-invasive, which is commonly used for the management of pain. It works via the application of electrical stimuli using adhesive gel pads. They are cheap to run and are widely accepted by patients. Hence application of TENS over acupoints (Acu-TENS) may provide a novel non-invasive treatment.

A randomised controlled trial will be carried out on patients with FI. Demographic data, past medical history, in particular any structural or neurological causes of FI, will be recorded. Ano-rectal manometry and endoanal ultrasound will be performed before and after treatment. Acu-TENS machine will be applied to standardised acupuncture points. Assessment of FI via Cleveland Clinic Florida Faecal Incontinence Score and Quality of life measurements via the validated questionnaires Short Form 36 (SF-36) and the Fecal Incontinence Quality of Life Scale (FIQL) (Chinese version) questionnaires will be carried out at baseline, and followup intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Acupuncture naïve patients
* Faecal incontinence with solid or liquid stool causing disruption of lifestyle
* Psychological stability and suitability as determined by the investigator
* Failed conservative or surgical treatment
* Intact peripheral neurosensory nervous system as determined by clinical investigation
* Able to read and write

Exclusion Criteria:

* Major internal and/or external sphincter defect (>120 degrees of sphincter circumference)
* Faecal impaction
* Presence of full thickness rectal prolapse
* Patients who have contact allergies to adhesive pads
* Implanted pacemaker, defibrillator, cardiopathy
* Pregnancy or intention to become pregnant
* Neurogenic or congenital disorders resulting in faecal incontinence (e.g. Multiple Sclerosis, uncontrolled diabetes, Parkinson's disease, Spina Bifida)
* Inflammatory bowel disease
* Chronic diarrhoea uncontrolled by medication or diet
* Previous rectal surgery (rectopexy or rectal resection)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of AcuTENS as treatment for faecal incontinence compared with sham intervention | post treatment 8 weeks and 6 months compared with baseline
  Response to treatment is defined as 50% or greater change in Faecal incontinence Severity index score compared to sham

SECONDARY OUTCOMES:
Changes in the severity of faecal incontience | post treatment 8 weeks and 6 months compared with baseline
  Wexner score will be used the assess the severity of faecal incontinence
Episodes of faecal urgency per week | post treatment 8 weeks and 6 months compared with baseline
  the number of episodes of faecal urgency experienced by the patient per week
Reduction in the number of incontinence episode per week | post treatment 8 weeks and 6 months compared with baseline
  the number of episodes of faecal incontience experienced by the patient per week
Differences in Quality of Life score between two groups | post treatment 8 weeks and 6 months compared with baseline
  using the tradition chinese version of the faecal incontinence quality of life questionnaire (FIQL)

CONTACTS AND LOCATIONS:
Overall Officials: Tony WC Mak, MD, FRCS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No